CLINICAL TRIAL: NCT01760031
Title: Remote Preconditioning for Contrast-Induced Acute Kidney Injury: Long-Term Follow up (RenPro Longterm)
Brief Title: Longterm Follow-up After Remote Ischemic Preconditioning for Prevention of Contrast-induced Nephropathy
Acronym: RenProLong
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Fikret Er, Assistant Professor, University of Cologne
Other Study IDs: RenPro1L
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Impaired Renal Function
Keywords: preconditioning; contrast-induced acute kidney injury; renal faliure
MeSH Terms: conditions — Renal Insufficiency | interventions — Ischemic Preconditioning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects with impaired renal function: Subjects with baseline impaired renal function undergoing cardiac catheterization with contrast-medium exposure
  Interventions: Other: Ischemic preconditioning

INTERVENTIONS:
Other: Ischemic preconditioning — Subjects received ischemic preconditioning previous to cardiac catheterization

SUMMARY:
Remote ischemic preconditioning reduces the incidence of contrast-induced acute kidney injury in patients undergoing elective coronary angiography. This study was designed to acquire long-term data of initially randomized patients in the RenPro Trial.

DETAILED DESCRIPTION:
Data of the RenPro Trial has been already published. In the present study data of longterm follow up are collected.

ELIGIBILITY:
All patients who participated to the RenPro trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients refered for elective cardiac catherization to the university hospital of Cologne. All patients who participated to the RenPro trial (www.germanctr.de; DRKS-ID DRKS00000666)
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
MACCE | 1 Year
  Major Adverse Cardiac and Cerebrovascular Events (Combined primary endpoint):
  All-cause mortality, cardiovascular mortality, rehospitalization, stroke, myocardial infarction, hemodialysis

SECONDARY OUTCOMES:
Renal function | 1 year
  changes of serum creatinine, eGFR, NGAL and cystatin C compared to baseline in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fikret Er, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Er F, Nia AM, Dopp H, Hellmich M, Dahlem KM, Caglayan E, Kubacki T, Benzing T, Erdmann E, Burst V, Gassanov N. Ischemic preconditioning for prevention of contrast medium-induced nephropathy: randomized pilot RenPro Trial (Renal Protection Trial). Circulation. 2012 Jul 17;126(3):296-303. doi: 10.1161/CIRCULATIONAHA.112.096370. Epub 2012 Jun 26. PMID 22735306